CLINICAL TRIAL: NCT04962178
Title: A Randomized Multicenter Trial to Evaluate Early Invasive Strategy for Patients With Acute ST-segment Elevation Myocardial Infarction Presenting 24-48 Hours From Symptom Onset
Brief Title: Evaluate Early Invasive Strategy for Patients With STEMI Presenting 24-48 Hours From Symptom Onset
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZS AMI 24-48
Record Dates: First submitted 2021-06-23; First posted 2021-07-14 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI)
Keywords: ST-segment Elevation Myocardial Infarction (STEMI); Early Invasive Strategy
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Invasive Strategy (Experimental): Procedure: Primary PCI
  Interventions: Procedure: Primary PCI
- Conservative Strategy (Active Comparator): Procedure: Optimal medical therapy with primary PCI not performed.
  Interventions: Other: Optimal medical therapy with primary PCI not performed

INTERVENTIONS:
Procedure: Primary PCI — The patients assigned to early invasive strategy group will receive the primary PCI.
  Arms: Early Invasive Strategy
Other: Optimal medical therapy with primary PCI not performed — The patients assigned to conservative strategy group will receive optimal medical therapy before primary endpoint accomplished.
  Arms: Conservative Strategy

SUMMARY:
The primary objective of the trial is to evaluate the efficacy of early invasive strategy for STEMI patients within 24-48h of symptom onset.

DETAILED DESCRIPTION:
At present, timely primary percutaneous coronary intervention (PCI) is the preferred strategy for ST-segment elevation myocardial infarction (STEMI) patients within 24h of symptom onset. In stable STEMI patients presenting 12 to 48 hours from symptom onset, BRAVE-2 Trial (n = 365) showed improved myocardial salvage and 4-year survival in patients treated with primary PCI compared with conservative treatment alone. However, data is scarce about the reperfusion strategy focusing on STEMI patients within 24-48h of symptom onset. Further investigations are warranted to explore the best timing of invasive strategy for STEMI patients within 24-48h of symptom onset.

Given that no randomized clinical trial is designed especially for STEMI patients within 24-48h of symptom onset, and limited data is available to evaluate the efficacy of early invasive strategy for the special subgroup of STEMI patients, investigators plan to perform a controlled, randomized trial to evaluate the efficacy of early invasive strategy for STEMI patients within 24-48h of symptom onset.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 or over and less than 75 years old;
2. ECG: a) ≥2 mm ST-segment elevation in 2 contiguous precordial leads or ≥1 mm ST-segment elevation in 2 contiguous extremity leads; or b) new or presumable new left bundle branch block in the presence of typical symptoms;
3. Patents with STEMI with symptom onset between 24 and 48 hours before randomization;
4. Signed informed consent form prior to trial participation.

Exclusion Criteria:

1. Patents with STEMI with symptom onset <24h or >48h or uncertain time onset.
2. Prior administration of thrombolytic therapy or attempted PCI before randomization;
3. Presence of indications for primary PCI, such as persistent chest pain, cardiogenic shock, life-threatening arrhythmias or cardiac arrest, severe acute heart failure, and mechanical complications;
4. Coagulopathy, active peptic ulcer, history of cerebral or subarachnoid hemorrhage, stroke within 6 months, other contraindications for antiplatelet or anticoagulant therapy;
5. Known intolerance to antiplatelet (e.g. aspirin, clopidogrel, ticagrelor) and anticoagulant therapy (e.g. heparin, bivalirudin);
6. Presence of contraindications for CMR;
7. Congenital heart disease or severe valvular disease;
8. eGFR <30 ml/min/1.73 m2;
9. History of malignant tumors;
10. Combined with other diseases and life expectancy ≤12 months;
11. Pregnancy;
12. Inclusion in another clinical trial;
13. Inability to provide informed consent or not available for follow-up judged by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Myocardial infraction size assessed by cardiac magnetic resonance (CMR) | 7 days (from symptom onset)
  Late gadolinium enhancement (LGE) by CMR is performed for myocardial infarction size quantification.

SECONDARY OUTCOMES:
A composite of cardiac death, recurrent myocardial infarction, ischaemia-driven target vessel revascularization, and stoke | 30 days
Microvascular obstruction (MVO) assessed by CMR | 7 days (from symptom onset)
  Serial imaging sequence results from CMR.
Intramyocardial hemorrhage (IMH) assessed by CMR | 7 days (from symptom onset)
  Serial imaging sequence results from CMR.
Area at risk (AAR) assessed by CMR | 7 days (from symptom onset)
  Serial imaging sequence results from CMR.
Left ventricular ejection fraction (LVEF) assessed by CMR | 7 days (from symptom onset)
  Imaging parameters from CMR.
Left ventricular end-diastolic volume (LVEDV) assessed by CMR | 7 days (from symptom onset)
  Imaging parameters from CMR.
Left ventricular end-systolic volume (LVESV) assessed by CMR | 7 days (from symptom onset)
  Imaging parameters from CMR.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao W, Zhong X, Ma Y, Huang D, Wang R, Zhao S, Yang S, Qian J, Ge J. A randomized multicenter trial to evaluate early invasive strategy for patients with acute ST-segment elevation myocardial infarction presenting 24-48 hours from symptom onset: Protocol of the RESCUE-MI study. Am Heart J. 2022 Sep;251:54-60. doi: 10.1016/j.ahj.2022.05.002. Epub 2022 May 5. PMID 35525262